CLINICAL TRIAL: NCT01704261
Title: A Phase III, Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial to Study the Safety and Efficacy of the Addition of MK-3102 to Subjects With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Combination Therapy With Glimepiride and Metformin
Brief Title: Addition of Omarigliptin (MK-3102) to Participants With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Combination Therapy With Glimepiride and Metformin (MK-3102-022)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3102-022; 2012-002612-10 (EudraCT Number)
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Results first posted 2015-11-25 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 2-(2,5-difluorophenyl)-5-(2-(methylsulfonyl)-2,6-dihydropyrrolo(3,4-c)pyrazol-5(4H)-yl)tetrahydro-2H-pyran-3-amine; glimepiride; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omarigliptin (Experimental): Omarigliptin (MK-3102) 25 mg capsule administered orally once a week for 24 weeks. Participants continue pre-study concomitant therapy of open-label glimepiride tablet(s) orally once daily (total daily dose >=4 mg per day) and metformin tablet(s) orally once or twice daily (total daily dose >=1500 mg per day).
  Interventions: Drug: Omarigliptin; Drug: Glimepiride; Drug: Metformin
- Placebo (Placebo Comparator): Matching placebo to omarigliptin capsule administered orally once a week for 24 weeks. Participants continue pre-study concomitant therapy of open-label glimepiride tablet(s) orally once daily (total daily dose >=4 mg per day) and metformin tablet(s) orally once or twice daily (total daily dose >=1500 mg per day).
  Interventions: Drug: Matching placebo to Omarigliptin; Drug: Glimepiride; Drug: Metformin

INTERVENTIONS:
Drug: Omarigliptin — Omarigliptin 25 mg capsule administered orally once a week
  Arms: Omarigliptin
Drug: Matching placebo to Omarigliptin — Matching placebo to omarigliptin capsule administered orally once a week
  Arms: Placebo
Drug: Glimepiride — Open-label glimepiride tablet(s) administered orally once daily for a total daily dose >=4 mg. In the event of hypoglycemia, the glimepiride dose may be down-titrated to a minimum dose of 1 mg daily.
  Other Names: Amaryl®; Glimy
Drug: Metformin — Open-label metformin tablet(s) administered orally once or twice daily for a total daily dose >=1500 mg
  Other Names: Fortamet®; Glucophage®; Glucophage® XR; Glumetza®; Riomet®

SUMMARY:
This study will examine the safety and efficacy of the addition of omarigliptin in participants with type 2 diabetes mellitus with inadequate glycemic control on metformin and glimepiride. The primary hypothesis is that after 24 weeks, the addition of treatment with omarigliptin provides a greater reduction in hemoglobin A1c (A1C) compared with the addition of placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes mellitus
* Currently taking stable doses of metformin (>=1500 mg/day) and sulfonylurea
* Male, or female not of reproductive potential or female of reproductive potential who agrees to remain abstinent or use (or have their partner use) 2 methods of acceptable contraception to prevent pregnancy during the study and for 21 days after the last dose of study drug

Exclusion Criteria:

* History of type 1 diabetes mellitus or a history of ketoacidosis
* Treated with any antihyperglycemic agent therapies other than the protocol-required sulfonylurea and metformin within 12 weeks prior to study participation or with omarigliptin at any time prior to study participation.
* History of hypersensitivity to a dipeptidyl peptidase IV (DPP-4) inhibitor
* On a weight loss program and is not in the maintenance phase; or has been on a weight loss medication in the past 6 months; or has undergone bariatric surgery within 12 months prior to study participation.
* Is on or likely to require treatment for >=2 consecutive weeks or repeated courses of corticosteroids (inhaled, nasal or topical corticosteroids are permitted)
* Currently being treated for hyperthyroidism or is on thyroid replacement therapy and has not been on a stable dose for at least 6 weeks
* Medical history of active liver disease (other than non-alcoholic hepatic steatosis), including chronic active hepatitis B or C, primary biliary cirrhosis, or symptomatic gallbladder disease
* Human immunodeficiency virus (HIV)
* New or worsening coronary heart disease, congestive heart failure, myocardial infarction, unstable angina, coronary artery intervention, stroke, or transient ischemic neurological disorder within the past 3 months
* Poorly controlled hypertension
* History of malignancy <=5 years prior to study participation, except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer
* Clinically important hematological disorder (such as aplastic anemia, myeloproliferative or myelodysplastic syndromes, thrombocytopenia)
* Pregnant or breast feeding, or is expecting to conceive or donate eggs during the trial, including 21 days following the last dose of study drug
* Current user of recreational or illicit drugs or has had a recent history of drug abuse or routinely consumes >2 alcoholic drinks per day or >14 drinks per week, or engages in binge drinking
* Donated blood products within 8 weeks of study participation, or intends to donate blood products during the study or has received or anticipates receiving blood products within 12 weeks prior to study participation or during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2012-10-18 (Actual); Primary Completion 2014-12-23 (Actual); Study Completion 2014-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Lee SH, Gantz I, Round E, Latham M, O'Neill EA, Ceesay P, Suryawanshi S, Kaufman KD, Engel SS, Lai E. A randomized, placebo-controlled clinical trial evaluating the safety and efficacy of the once-weekly DPP-4 inhibitor omarigliptin in patients with type 2 diabetes mellitus inadequately controlled by glimepiride and metformin. BMC Endocr Disord. 2017 Nov 6;17(1):70. doi: 10.1186/s12902-017-0219-x. PMID 29110647
- Available data/document: CSR Synopsis Links — http://www.merck.com/clinical-trials/study.html?id=3102-022&kw=3102-022&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty-one sites received IEC/IRB approval and were shipped clinical supplies.
Pre-assignment Details: In total, 583 participants were screened and 276 participants were excluded during screening. The most common reason for participants not being randomized was screen failure. The most common reasons for screen failure were not meeting the metformin and glimepiride dose requirements inclusion criterion or meeting exclusionary laboratory values.
Groups:
- Omarigliptin: Omarigliptin 25 mg capsule administered orally once a week for 24 weeks. Participants continue pre-study concomitant therapy of open-label glimepiride tablet(s) orally once daily (total daily dose >=4 mg per day) and metformin tablet(s) orally once or twice daily (total daily dose >=1500 mg per day).
Period: Overall Study
Arm/Group | Omarigliptin | Placebo
Started | 154 | 153
Completed | 141 | 138
Not Completed | 13 | 15
Not completed — Withdrawal by Subject | 12 | 15
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omarigliptin | Placebo | Total
Number analyzed (Participants) | 154 | 153 | 307
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.2 (8.4) | 58.4 (9.4) | 57.8 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 79 | 160
  Male | 73 | 74 | 147

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (A1C) at Week 24
Description: A1C is blood marker used to report average blood glucose levels over a prolonged periods of time and is reported as a percentage (%). Thus, this change from baseline reflects the Week 24 A1C minus the Week 0 A1C.
Time Frame: Baseline and Week 24
Population: The Full Analysis Set (FAS) population consisted of all randomized participants who received at least 1 dose of study medication and had a baseline measurement or a measurement for the analysis endpoint after receiving study medication. One participant was in 2 clinical trials in parallel and was excluded from all efficacy and safety analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: %A1C
Arm/Group | Omarigliptin | Placebo
Number analyzed (Participants) | 153 | 153
%A1C | -0.67 [-0.84 to -0.50] | -0.06 [-0.23 to 0.12]
Statistical Analysis 1: Comparison: Omarigliptin vs Placebo; Test type: Superiority or Other; p < 0.001, Difference in the least squares means; Based on a constrained longitudinal data analysis (cLDA) method with a restriction of the same baseline mean across treatment groups; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-0.85 to -0.38]

2. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure.
Time Frame: Up to Week 27
Population: All Subjects as Treated (ASaT) population, defined as all randomized participants who received at least 1 dose of study medication. Participants were included in the treatment group corresponding to the study treatment they actually received. One participant was in 2 clinical trials and was excluded from all efficacy and safety analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin | Placebo
Number analyzed (Participants) | 153 | 153
Percentage of participants | 57.5 | 47.7
Statistical Analysis 1: Comparison: Omarigliptin vs Placebo; Test type: Superiority or Other; Difference in % Omarigliptin vs Placebo = 9.8, 95% CI 2-sided [-1.4 to 20.8]

3. Primary Outcome: Percentage of Participants Who Discontinued From the Study Due to an AE
Description: as for outcome 2
Time Frame: Up to Week 24
Population: The ASaT Population was defined as all randomized participants who received at least 1 dose of study medication. Participants were included in the treatment group corresponding to the study treatment they actually received. One participant was in 2 clinical trials and was excluded from all efficacy and safety analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin | Placebo
Number analyzed (Participants) | 153 | 153
Percentage of participants | 2.6 | 2.6
Statistical Analysis 1: Comparison: Omarigliptin vs Placebo; Test type: Superiority or Other; Difference in % Omarigliptin vs Placebo = 0, 95% CI 2-sided [-4.3 to 4.3]

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Blood glucose was measured on a fasting basis. FPG is expressed as mg/dL. Blood was drawn at predose on Day 1 and after 24 weeks of treatment to determine change in plasma glucose levels (i.e., FPG at Week 24 minus FPG at baseline).
Time Frame: Baseline and Week 24
Population: The FAS population consisted of all randomized participants who received at least 1 dose of study medication and had a baseline measurement or a measurement for the analysis endpoint after receiving study medication. One participant was in 2 clinical trials in parallel and was excluded from all efficacy and safety analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin | Placebo
Number analyzed (Participants) | 153 | 153
mg/dL | -19.6 [-26.7 to -12.5] | -3.0 [-10.2 to 4.1]
Statistical Analysis 1: Comparison: Omarigliptin vs Placebo; Test type: Superiority or Other; p < 0.001, Difference in the least squares means; [statistical method as in outcome 1, analysis 1]; Difference of the least squares means = -16.6, 95% CI 2-sided [-25.5 to -7.8]

5. Secondary Outcome: Percentage of Participants Attaining A1C Glycemic Goals of <7% and <6.5% at Week 24
Description: The percentage of participants who achieved A1C values <6.5% (48 mmol/mol) or <7.0% (53 mmol/mol) in the FAS population at Week 24.
Time Frame: 24 weeks
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Omarigliptin | Placebo
Number analyzed (Participants) | 153 | 153
Percentage of participants
  <7.0% | 23.8 [17.5 to 31.5] | 4.4 [2.1 to 9.3]
  <6.5% | 10.1 [6.1 to 16.4] | 2.1 [0.7 to 6.0]
Statistical Analysis 1: Comparison: Omarigliptin vs Placebo; Test type: Superiority or Other; p < 0.001, Miettinen & Nurminen method; Between-group confidence intervals and p-value (%) A1C <7.0%; estimated using standard multiple imputation techniques; Between-group Rate Difference = 19.3, 95% CI 2-sided [11.7 to 27.6]
Statistical Analysis 2: Comparison: Omarigliptin vs Placebo; Test type: Superiority or Other; p = 0.005, Miettinen & Nurminen method; Between-group confidence intervals and p-value (%) A1C <7.0%; estimated using standard multiple imputation techniques; Between-group Rate Difference (%) = 8.0, 95% CI 2-sided [2.7 to 14.5]

ADVERSE EVENTS:
Time Frame: Up to Week 27
Description: The ASaT Population was all randomized participants who received at least one study drug. Participants were included in the treatment group corresponding to the study treatment they actually received. One participant was in 2 clinical trials and was excluded from all efficacy and safety analysis.
Arm/Group | Omarigliptin | Placebo
Serious Adverse Events (participants affected / at risk) | 3/153 | 5/153
Other Adverse Events (participants affected / at risk) | 29/153 | 23/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin (N=153) | Placebo (N=153)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin (N=153) | Placebo (N=153)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 9 (11)
Urinary tract infection (Infections and infestations) | 9 (9) | 3 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 18 (65) | 13 (44)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.